CLINICAL TRIAL: NCT02784444
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, 12-Month, Multiple-Dose Study to Evaluate the Safety, Tolerability and Efficacy of Three Dose Levels of MSDC-0602K in Patients With NASH (EMMINENCE™)
Brief Title: A Study to Evaluate the Safety, Tolerability & Efficacy of MSDC-0602K in Patients With NASH
Acronym: EMMINENCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cirius Therapeutics, Inc. (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSDC-0602K-C009NASH
Record Dates: First submitted 2016-05-18; First posted 2016-05-27 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Non-alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis; NASH - Nonalcoholic Steatohepatitis
Keywords: NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- MSDC-0602K Dose 1 capsules (Active Comparator): MSDC-0602K Dose 1 capsule taken once daily for 360 days
  Interventions: Drug: MSDC-0602K
- MSDC-0602K Dose 2 capsules (Active Comparator): MSDC-0602K Dose 2 capsules taken once daily for 360 days
  Interventions: Drug: MSDC-0602K
- MSDC-0602K Dose 3 capsules (Active Comparator): MSDC-0602K Dose 3 capsules taken once daily for 360 days
  Interventions: Drug: MSDC-0602K
- Placebo capsules (Placebo Comparator): Matching Placebo capsule taken once daily for 360 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MSDC-0602K — MSDC-0602K capsules
  Arms: MSDC-0602K Dose 1 capsules; MSDC-0602K Dose 2 capsules; MSDC-0602K Dose 3 capsules
Drug: Placebo — Placebo capsules
  Arms: Placebo capsules

SUMMARY:
This is a randomized, double-blinded study of three doses of MSDC-0602K or placebo given orally once daily to subjects with biopsy proven NASH with fibrosis and no cirrhosis.

DETAILED DESCRIPTION:
This is a randomized, double-blinded study of three doses of MSDC-0602K or placebo given orally once daily to subjects with biopsy proven NASH with fibrosis and no cirrhosis. Visits to the clinic will be at baseline, 1, 2, 3, 6, 9, and 12 months, with one 2- week follow-up visit.

Safety will be assessed by monitoring of vital signs, 12 lead electrocardiogram (ECG), physical examinations, safety labs, and adverse events (AEs).

ELIGIBILITY:
Selected Inclusion Criteria:

* Adult subjects 18 years of age or greater
* Histological evidence of NASH, based on biopsy, with a NAS (NASH CRN scoring) ≥ 4 with a score of at least 1 in each component of NAS.
* Histological evidence of liver fibrosis defined as NASH CRN System fibrosis score F1 to F3.
* Subjects with type 2 diabetes mellitus (DM) must be under stable and reasonable control.
* Male and female subjects who are taking Vitamin E should be on a stable dose of Vitamin E (if ≥ 400 IU) for a period of at least 3 months prior to randomization.
* Females should be either postmenopausal (at least 12 months since last menses) or surgically sterilized (bilateral tubal ligation or hysterectomy). Males with female partners of child-bearing potential must agree to use adequate contraceptive methods (including a condom, plus one other form of contraception) if engaging in sexual intercourse.
* Willing and able to sign an informed consent document indicating understanding the purpose of and procedures required for the study and willingness to participate in the study.

Selected Exclusion Criteria:

* Known history of HIV.
* Prior liver transplantation.
* Other well-documented causes of active chronic liver disease.
* History of cirrhosis and/or hepatic decompensation including ascites, hepatic encephalopathy or variceal bleeding.
* History of alcohol abuse or drug abuse within 6 months of Screening.
* Type 1 diabetes mellitus.
* Current or history of recent (≤ 6 months) use of ursodeoxycholic acid.
* Use of concomitant medications with a known significant metabolism by CYP2C8 or CPY2C9.
* History of diabetic ketoacidosis or hyperosmolar non-ketotic coma within 6 months prior to randomization.
* History of heart failure (including CHF) or previous cardiovascular event (myocardial infarct, by-pass surgery, or PTCA) within the past 6 months prior to randomization.
* Blood pressure greater than 160/100 mmHg.
* Participation in an investigational study or received an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to study drug administration.
* Malignancy, including leukemia and lymphoma (excluding basal cell and squamous skin cell cancers and localized prostrate cancer) treated within the last 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Dittrich, MD, Study Director — Cirius Therapeutics, Inc.
Locations (40):
- United States (40):
  - Chandler, Arizona
  - Tucson, Arizona
  - Chula Vista, California
  - Fresno, California
  - Garden Grove, California
  - Huntington Park, California
  - La Mesa, California
  - Los Angeles, California
  - Poway, California
  - Rialto, California
  - San Diego, California
  - Englewood, Colorado
  - Gainesville, Florida
  - Hialeah, Florida
  - Inverness, Florida
  - Lakewood Rch, Florida
  - Miami Lakes, Florida
  - Wellington, Florida
  - Marietta, Georgia
  - Indianapolis, Indiana
  - Bastrop, Louisiana
  - New Orleans, Louisiana
  - West Monroe, Louisiana
  - Flowood, Mississippi
  - Brooklyn, New York
  - New York, New York
  - Fayetteville, North Carolina
  - Greenville, North Carolina
  - Statesville, North Carolina
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Hermitage, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - Fort Sam Houston, Texas
  - Houston, Texas
  - Live Oak, Texas
  - Rollingwood, Texas
  - San Antonio, Texas
  - Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harrison SA, Alkhouri N, Davison BA, Sanyal A, Edwards C, Colca JR, Lee BH, Loomba R, Cusi K, Kolterman O, Cotter G, Dittrich HC. Insulin sensitizer MSDC-0602K in non-alcoholic steatohepatitis: A randomized, double-blind, placebo-controlled phase IIb study. J Hepatol. 2020 Apr;72(4):613-626. doi: 10.1016/j.jhep.2019.10.023. Epub 2019 Nov 4. PMID 31697972

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching Placebo capsule taken once daily for 360 days
  Placebo: Placebo capsules
- MSDC-0602K 62.5 mg: MSDC-0602K 62.5 mg taken once daily for 360 days
  MSDC-0602K: MSDC-0602K capsules
- MSDC-0602K 125 mg: MSDC-0602K 125 mg taken once daily for 360 days
  MSDC-0602K: MSDC-0602K capsules
- MSDC-0602K 250 mg: MSDC-0602K 250 mg taken once daily for 360 days
  MSDC-0602K: MSDC-0602K capsules
Period: Overall Study
Arm/Group | Placebo | MSDC-0602K 62.5 mg | MSDC-0602K 125 mg | MSDC-0602K 250 mg
Started | 94 | 99 | 98 | 101
Completed | 78 | 90 | 86 | 88
Not Completed | 16 | 9 | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MSDC-0602K 62.5 mg | MSDC-0602K 125 mg | MSDC-0602K 250 mg | Total
Number analyzed (Participants) | 94 | 99 | 98 | 101 | 392
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (11.2) | 56.9 (10.3) | 56.0 (10.9) | 56.8 (10.4) | 56.1 (10.64)
Age, Customized [Count of Participants; unit: Participants]
  Age at Enrollment: < 55 years | 43 | 35 | 42 | 37 | 157
  Age at Enrollment: >= 55 years | 51 | 64 | 56 | 64 | 235
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 56 | 63 | 58 | 228
  Male | 43 | 43 | 35 | 43 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 32 | 29 | 33 | 119
  Not Hispanic or Latino | 69 | 67 | 69 | 68 | 273
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian Or Alaska Native | 0 | 0 | 1 | 0 | 1
  Race: Asian | 2 | 2 | 2 | 2 | 8
  Race: Black Or African American | 5 | 3 | 3 | 3 | 14
  Race: Native Hawaiian Or Other Pacific Islander | 0 | 0 | 1 | 2 | 3
  Race: Other | 2 | 1 | 0 | 3 | 6
  Race: White | 85 | 93 | 91 | 91 | 360

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hepatic Histological Improvement in NAS
Description: * A decrease of at least 2 points in NAS at 12 months.
  * At least a 1 point reduction in either ballooning or inflammation from baseline to 12 months.
  * no increase in CRN fibrosis score (i.e., an increase of 1 stage or more) from baseline to 12 months.
Time Frame: 12 months (360 days)
Population: Subjects in the Modified Intent-to-Treat Set with available baseline biopsy and 12-month biopsy taken within 14 days of study drug discontinuation.
Measure: Number; unit: Participants
Arm/Group | Placebo | MSDC-0602K 62.5 mg | MSDC-0602K 125 mg | MSDC-0602K 250 mg
Number analyzed (Participants) | 74 | 84 | 82 | 86
Participants | 22 | 25 | 27 | 34
Statistical Analysis 1: Comparison: Placebo vs MSDC-0602K 62.5 mg; The null hypothesis is that there is no difference in response rates between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.747, Regression, Logistic — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Models are adjusted for presence of diabetes mellitus, baseline fibrosis F1 versus F2/F3, and baseline NAS (0-8); Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.44 to 1.81]
Statistical Analysis 2: Comparison: Placebo vs MSDC-0602K 125 mg; The null hypothesis is that there is no difference in response rates between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.575, Regression, Logistic — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Models are adjusted for presence of diabetes mellitus, baseline fibrosis F1 versus F2/F3, and baseline NAS (0-8); Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.60 to 2.48]
Statistical Analysis 3: Comparison: Placebo vs MSDC-0602K 250 mg; The null hypothesis is that there is no difference in response rates between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.158, Regression, Logistic — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Models are adjusted for presence of diabetes mellitus, baseline fibrosis F1 versus F2/F3, and baseline NAS (0-8); Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.83 to 3.27]

2. Secondary Outcome: Number of Subjects With Resolution of NASH With no Worsening of Fibrosis at 12 Months.
Description: * CRN ballooning score of 0 at 12-months
  * CRN inflammation score of 0 or 1 at 12-months
  * No increase in CRN fibrosis score from baseline to 12-months
Time Frame: 12 months (360 days)
Population: Analysis Population Description: Subjects in the Modified Intent-to-Treat Set with available baseline biopsy and 12-month biopsy taken within 14 days of study drug discontinuation.
Measure: Number; unit: Participants
Arm/Group | Placebo | MSDC-0602K 62.5 mg | MSDC-0602K 125 mg | MSDC-0602K 250 mg
Number analyzed (Participants) | 74 | 84 | 82 | 86
Participants | 15 | 17 | 23 | 27
Statistical Analysis 1: Comparison: Placebo vs MSDC-0602K 62.5 mg; The null hypothesis is that there is no difference in response rates between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.828, Regression, Logistic — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Models are adjusted for presence of diabetes mellitus, baseline fibrosis F1 versus F2/F3, and baseline NAS (0-8); Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.49 to 2.42]
Statistical Analysis 2: Comparison: Placebo vs MSDC-0602K 125 mg; The null hypothesis is that there is no difference in response rates between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.299, Regression, Logistic — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Models are adjusted for presence of diabetes mellitus, baseline fibrosis F1 versus F2/F3, and baseline NAS (0-8); Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.70 to 3.21]
Statistical Analysis 3: Comparison: Placebo vs MSDC-0602K 250 mg; The null hypothesis is that there is no difference in response rates between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.116, Regression, Logistic — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Models are adjusted for presence of diabetes mellitus, baseline fibrosis F1 versus F2/F3, and baseline NAS (0-8); Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.86 to 3.82]

3. Secondary Outcome: Number of Subjects With Improvement of Fibrosis (CRN Staging Score) by at Least 1 Stage With no Worsening of NASH at 12 Months.
Description: * Decrease in fibrosis CRN staging score of >= 1 full stage from baseline to 12 months
  * No increase in ballooning CRN score from baseline to 12 months
  * No increase in inflammation CRN score from baseline to 12-months
Time Frame: 12 months (360 days)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | MSDC-0602K 62.5 mg | MSDC-0602K 125 mg | MSDC-0602K 250 mg
Number analyzed (Participants) | 74 | 84 | 82 | 86
Participants | 16 | 20 | 23 | 25
Statistical Analysis 1: Comparison: Placebo vs MSDC-0602K 62.5 mg; The null hypothesis is that there is no difference in response rates between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.657, Regression, Logistic — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Models are adjusted for presence of diabetes mellitus, baseline fibrosis F1 versus F2/F3, and baseline NAS (0-8); Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.55 to 2.55]
Statistical Analysis 2: Comparison: Placebo vs MSDC-0602K 125 mg; The null hypothesis is that there is no difference in response rates between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.332, Regression, Logistic — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Models are adjusted for presence of diabetes mellitus, baseline fibrosis F1 versus F2/F3, and baseline NAS (0-8); Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.69 to 3.06]
Statistical Analysis 3: Comparison: Placebo vs MSDC-0602K 250 mg; The null hypothesis is that there is no difference in response rates between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.270, Regression, Logistic — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Models are adjusted for presence of diabetes mellitus, baseline fibrosis F1 versus F2/F3, and baseline NAS (0-8); Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.72 to 3.16]

4. Secondary Outcome: Mean Change From Baseline in NAFLD Activity Score (NAS)
Description: NAS is the sum of the scores of steatosis, inflammation, and ballooning. It has a range of 0 to 8 with higher scores indicating worse disease severity.
Time Frame: 12 months (360 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | MSDC-0602K 62.5 mg | MSDC-0602K 125 mg | MSDC-0602K 250 mg
Number analyzed (Participants) | 74 | 84 | 83 | 86
Scores on a scale | -0.6 (1.80) | -1.0 (1.66) | -1.1 (1.74) | -1.2 (1.83)
Statistical Analysis 1: Comparison: Placebo vs MSDC-0602K 62.5 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.392, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Model adjusted by age, sex, presence of diabetes mellitus, Vitamin E ≥ 400 IU, baseline fibrosis F1 versus F2/F3, and baseline NAS (0-8); Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.7 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs MSDC-0602K 125 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.023, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.1 to -0.1]
Statistical Analysis 3: Comparison: Placebo vs MSDC-0602K 250 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.028, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.0 to -0.1]

5. Secondary Outcome: Mean Change From Baseline in CRN Steatosis Score
Description: Steatosis is assessed on a scale of 0 to 3 with higher scores indicating more severe steatosis.
Time Frame: 12 months (360 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | MSDC-0602K 62.5 mg | MSDC-0602K 125 mg | MSDC-0602K 250 mg
Number analyzed (Participants) | 74 | 84 | 83 | 86
Scores on a scale | -0.4 (0.80) | -0.6 (0.88) | -0.5 (0.93) | -0.7 (0.94)
Statistical Analysis 1: Comparison: Placebo vs MSDC-0602K 62.5 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.224, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Model adjusted by age, sex, presence of diabetes mellitus, Vitamin E ≥ 400 IU, baseline fibrosis F1 versus F2/F3, and baseline steatosis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs MSDC-0602K 125 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.096, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0]
Statistical Analysis 3: Comparison: Placebo vs MSDC-0602K 250 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.007, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to -0.1]

6. Secondary Outcome: Mean Change From Baseline in CRN Inflammation Score
Description: Inflammation is assessed on a scale of 0 to 3 with higher scores indicating more severe inflammation.
Time Frame: 12 months (360 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | MSDC-0602K 62.5 mg | MSDC-0602K 125 mg | MSDC-0602K 250 mg
Number analyzed (Participants) | 74 | 84 | 83 | 86
Scores on a scale | -0.1 (0.70) | -0.1 (0.71) | -0.2 (0.56) | -0.1 (0.66)
Statistical Analysis 1: Comparison: Placebo vs MSDC-0602K 62.5 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.488, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Model adjusted by age, sex, presence of diabetes mellitus, Vitamin E ≥ 400 IU, baseline fibrosis F1 versus F2/F3, and baseline inflammation; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs MSDC-0602K 125 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.291, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs MSDC-0602K 250 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.595, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.1]

7. Secondary Outcome: Mean Change From Baseline in CRN Ballooning Score
Description: Hepatocellular ballooning is assessed on a scale of 0 to 2 with higher scores indicating more severe hepatocellular ballooning.
Time Frame: 12 months (360 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | MSDC-0602K 62.5 mg | MSDC-0602K 125 mg | MSDC-0602K 250 mg
Number analyzed (Participants) | 74 | 84 | 83 | 86
Scores on a scale | -0.2 (0.98) | -0.4 (0.94) | -0.4 (0.94) | -0.4 (0.91)
Statistical Analysis 1: Comparison: Placebo vs MSDC-0602K 62.5 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.416, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Model adjusted by age, sex, presence of diabetes mellitus, Vitamin E ≥ 400 IU, baseline fibrosis F1 versus F2/F3, and baseline ballooning; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs MSDC-0602K 125 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.056, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to 0.0]
Statistical Analysis 3: Comparison: Placebo vs MSDC-0602K 250 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.220, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.1]

8. Secondary Outcome: Mean Change From Baseline in CRN Fibrosis Staging Score
Description: Fibrosis is assessed on a scale of 0 to 4 with higher scores indicating more severe fibrosis.
Time Frame: 12 months (360 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | MSDC-0602K 62.5 mg | MSDC-0602K 125 mg | MSDC-0602K 250 mg
Number analyzed (Participants) | 74 | 84 | 82 | 86
Scores on a scale | 0.0 (1.10) | 0.1 (1.07) | -0.1 (1.16) | -0.1 (1.27)
Statistical Analysis 1: Comparison: Placebo vs MSDC-0602K 62.5 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.928, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; Model adjusted by age, sex, diabetes mellitus, Vitamin E ≥ 400 IU, baseline fibrosis F1 vs. F2/F3, and baseline CRN fibrosis staging score; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs MSDC-0602K 125 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.244, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs MSDC-0602K 250 mg; The null hypothesis is that there is no difference in changes between the MSDC-0602K dose and placebo; Test type: Superiority; p = 0.228, ANCOVA — Statistical testing was two-sided using a significance (alpha) level of 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to the final study visit, at an average of 1 year and 2 weeks.
Arm/Group | Placebo | MSDC-0602K 62.5 mg | MSDC-0602K 125 mg | MSDC-0602K 250 mg
All-Cause Mortality (participants affected / at risk) | 1/94 | 0/99 | 1/98 | 0/101
Serious Adverse Events (participants affected / at risk) | 9/94 | 5/99 | 13/98 | 7/101
Other Adverse Events (participants affected / at risk) | 75/94 | 78/99 | 76/98 | 77/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | MSDC-0602K 62.5 mg (N=99) | MSDC-0602K 125 mg (N=98) | MSDC-0602K 250 mg (N=101)
Diverticultis (Infections and infestations) | 1 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Urinary tract infections (Infections and infestations) | 0 | 1 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Brain stem ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Malignant hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Transurethral prostatetectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | MSDC-0602K 62.5 mg (N=99) | MSDC-0602K 125 mg (N=98) | MSDC-0602K 250 mg (N=101)
Urinary tract infection (Infections and infestations) | 4 | 10 | 3 | 5
Sinusitis (Infections and infestations) | 5 | 6 | 5 | 4
Influenza (Infections and infestations) | 0 | 5 | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 7 | 6 | 3 | 5
Bronchitis (Infections and infestations) | 3 | 2 | 6 | 5
Nausea (Gastrointestinal disorders) | 7 | 8 | 7 | 13
Dirrhoea (Gastrointestinal disorders) | 5 | 7 | 9 | 4
Constipation (Gastrointestinal disorders) | 5 | 7 | 5 | 7
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4 | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 4 | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 5 | 1 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 5 | 4
Procedural pain (Injury, poisoning and procedural complications) | 8 | 5 | 2 | 3
Oedema peripheral (General disorders) | 6 | 5 | 9 | 5
Headache (Nervous system disorders) | 2 | 4 | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 5 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT02784444/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT02784444/SAP_001.pdf